CLINICAL TRIAL: NCT01199926
Title: Impact of Vitamin D Supplementation on Strength and Lean Mass Accumulation During an Exercise Intervention
Brief Title: Effect of Vitamin D Supplementation on Muscle Mass and Function
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Purdue University (Other)
Responsible Party: Principal Investigator, Dorothy Teegarden, Associate Dean Research and Grad. Prof. College of HHS, Purdue University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: GSSI-VitD (0801006402)
Record Dates: First submitted 2010-09-09; First posted 2010-09-13 (Estimated); Results first posted 2015-05-15 (Estimated); Last update posted 2015-05-15 (Estimated); Status verified 2015-04

CONDITIONS: Obesity; Insulin Resistance; Inflammation
Keywords: 25-hydroxyvitamin D; Parathyroid hormone; Lean mass; Muscular strength; Glucose tolerance
MeSH Terms: conditions — Obesity; Insulin Resistance; Inflammation | interventions — Vitamin D; Cholecalciferol; microcrystalline cellulose

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitamin D (Experimental): Participants in this arm consumed a 4000 IU vitamin D supplement daily for 12 weeks while participating in a resistance exercise training program.
  Interventions: Dietary Supplement: Vitamin D
- Placebo (Placebo Comparator): Participants in this arm consumed a placebo (microcrystalline cellulose) daily for 12 weeks while participating in a resistance exercise training program.
  Interventions: Dietary Supplement: Vitamin D; Drug: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin D — 4000 IU of vitamin D per day for 12 weeks.
  Other Names: cholecalciferol
Drug: Placebo — Placebo (microcrystalline cellulose) ingestion each day for 12 weeks.
  Other Names: microcrystalline cellulose
  Arms: Placebo

SUMMARY:
The study was designed to assess the effects of vitamin D supplementation during exercise training on body composition, muscle function, and glucose tolerance. The investigators hypothesis for these studies is that vitamin D supplementation enhances exercise-induced increases in strength and lean mass, potentially through enhancing insulin sensitivity and reducing inflammation.

DETAILED DESCRIPTION:
The study was designed to assess the effects of vitamin D supplementation during exercise training on body composition, muscle function, and glucose tolerance. It was a double-blind, randomized, placebo-controlled, clinical trial with participants randomized into either a 4,000 IU/day vitamin D or placebo group and all participants completed 12 wks (3 d/wk) of exercise training.

ELIGIBILITY:
Inclusion Criteria:

* Physical activity scores in the "low" to "very low" category
* Fitness estimations in the "below average" or lower categories
* body mass index scores >24.9 indicating overweight or obesity.

Exclusion Criteria:

* Use of tanning booths or other artificial UV light exposure
* High baseline vitamin D and calcium intake
* Plans to visit sunny/warm destinations during the winter months/study period
* History or presence of metabolic disease, type 2 diabetes, eating disorders, gastrointestinal disorders, pregnancy or lactation
* Use of drugs to treat obesity (last 12 weeks)
* Use of over the counter anti-obesity agents (last 12 weeks)
* Recent initiation of an exercise program (last four weeks).

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2008-08; Primary Completion 2009-07 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dorothy Teegarden, PhD, Principal Investigator — Purdue University; Michael G Flynn, PhD, Principal Investigator — College of Charleston
Locations (1):
- Wastl Human Performance Laboratory, Purdue University, West Lafayette, Indiana, United States

REFERENCES:
- [Derived] Carrillo AE, Flynn MG, Pinkston C, Markofski MM, Jiang Y, Donkin SS, Teegarden D. Impact of vitamin D supplementation during a resistance training intervention on body composition, muscle function, and glucose tolerance in overweight and obese adults. Clin Nutr. 2013 Jun;32(3):375-81. doi: 10.1016/j.clnu.2012.08.014. Epub 2012 Aug 31. PMID 23034474

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Start Sept 2008 Recruitment at Purdue University
Pre-assignment Details: Following participant recruitment, baseline testing was completed prior to enrollment, study initiation and group assignment.
Groups:
- Vitamin D: Participants in this arm consumed a 4000 IU vitamin D3 supplement daily for 12 weeks while participating in a resistance exercise training program.
Period: Overall Study
Arm/Group | Vitamin D | Placebo
Started | 17 | 17
Completed | 10 | 13
Not Completed | 7 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vitamin D | Placebo | Total
Number analyzed (Participants) | 17 | 17 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 17 | 34
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 26 (4.5) | 26.2 (5.1) | 26.1 (4.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 7 | 7 | 14
Region of Enrollment [Number; unit: participants]
  United States | 17 | 17 | 34

OUTCOME MEASURES:

1. Primary Outcome: Muscle Function
Description: The primary endpoint is the change in lean mass (kilograms) after the three month resistance exercise intervention.
Time Frame: three months
Population: Power statistical calculation was completed based on 80% power and error on lean mass measurement.
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Vitamin D | Placebo
Number analyzed (Participants) | 10 | 13
kilograms | 1.14 (1.22) | 1.50 (1.16)

2. Primary Outcome: Glucose Tolerance
Description: The primary endpoint is the change in the area under the glucose curve following an oral glucose tolerance test prior to and after the three month intervention.
Time Frame: three months
Population: Power statistical calculation was completed based on 80% power and error on lean mass measurement.
Measure: Mean (Standard Deviation); unit: mmol/L/120 min
Arm/Group | Vitamin D | Placebo
Number analyzed (Participants) | 10 | 13
mmol/L/120 min | -18.0 (63.4) | -25.7 (31.1)

3. Primary Outcome: Inflammation
Description: The primary endpoint is the change in C reactive protein after the three month intervention
Time Frame: three months
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Vitamin D | Placebo
Number analyzed (Participants) | 10 | 13
mg/L | 0.64 (1.62) | -0.33 (2.60)

ADVERSE EVENTS:
Groups:
- Vitamin D: Were asked to consume 4000 IU of vitamin D/day for 3 months while performing a resistance training intervention.
- Placebo: Were asked to consume a placebo pill (microcrystalline cellulose) each day for 3 months while performing a resistance training intervention.
Arm/Group | Vitamin D | Placebo
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes